CLINICAL TRIAL: NCT03191435
Title: Effect of Inspiratory Muscle Training on Glycemic Control in Individuals With Type 2 Diabetes:Randomized Clinical Trial
Brief Title: Inspiratory Muscle Training on Glycemic Control in Individuals With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 61986916.9.0000.5327
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes mellitus, type 2; Inspiratory muscle training; Glycemic control; Glucose; Exercise; Diaphragm exercise; Inspiratory loading
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel Randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training (Experimental): Patients will perform the inspiratory muscle training using a load moderate of 30% of maximal inspiratory pressure (MIP 30%).
  Interventions: Device: Inspiratory muscle training.
- Placebo inspiratory muscle (Placebo Comparator): Patients will perform the inspiratory muscle training using a load of 2% of maximal inspiratory pressure (MIP 2%).
  Interventions: Device: Placebo inspiratory muscle

INTERVENTIONS:
Device: Inspiratory muscle training. — Patients will perform the inspiratory muscle training using a moderate load of 30% of maximal inspiratory pressure (MIP 30%). The training will be conducted at home in a period of 30 minutes, 7 times a week, during 12 weeks. During inspiratory muscle training, individuals will attend Hospital de Clinicas de Porto Alegre once a week to the supervision of the way the exercise is being performed. Furthermore, load in the device (powerbreathe) will be adjusted for the individual to use next week.
  Arms: Inspiratory muscle training
Device: Placebo inspiratory muscle — Patients will perform the inspiratory muscle training using a very low load of 2% of maximal inspiratory pressure (MIP 2%). The training will be conducted at home in a period of 30 minutes, 7 times a week, in the course of 12 weeks. During inspiratory muscle training, individuals will attend Hospital de Clinicas de Porto Alegre once a week to the supervision of the way the exercise is being performed.
  Arms: Placebo inspiratory muscle

SUMMARY:
In diabetic individuals, changes in ventilatory muscle strength and lung function have been demonstrated over the years. The onset and progression of chronic complications in diabetes should be avoided by reaching glycated hemoglobin (HbA1c) levels below 7%. The control of glycemia through the measurement of HbA1c is fundamental to avoid complications. The inspiratory muscle training has been used in several clinical situations, and may be an alternative for individuals with type 2 diabetes mellitus who have difficulties performing conventional exercises. The long-term effect of inspiratory muscle training on glycemic control has not been tested yet. The aim of this study is to evaluate the effects of inspiratory muscle training on glycemic control in individuals with type 2 diabetes.

DETAILED DESCRIPTION:
An acute high intensity inspiratory muscle exercise session was able to reduce glycemic levels (24%) similarly to an aerobic exercise session (25%) in subjects with type 2 diabetes, demonstrating that this type of exercise inspiratory muscle may have great potential in improving glycemic control.The present study will investigate if training of the inspiratory musculature for 8 and 12 weeks is capable of improving glycated hemoglobin, glucose and inspiratory muscle strength in individuals with type 2 diabetes. In addition, this study will evaluate the effect of inspiratory muscle training, with moderate loading of 30% of the MIP, on volumes and capacities lung in patients with type 2 diabetes. The subjects with type 2 diabetes will be recruited from the ambulatory of the Hospital de Clinicas de Porto Alegre and through newspaper advertisements.

Patients will be submitted to a general evaluation, including clinical history, physical examination, laboratory evaluation and application of the international physical activity questionnaire. Subsequently, individuals will perform assessments of lung functions (lung function assessment, ventilatory muscle strength test, inspiratory muscle strength test) and autonomic assessment (Ewing's tests). Patients will be randomized to perform inspiratory muscle training with a placebo load (MIP 2%) or with moderate intensity (MIP 30%). Upon the randomization, participants will initiate inspiratory musculature training. The exams of HbA1c, glucose and ventilatory muscle strength tests will be performed in three moments: 1) at the initial assessment, 2) in the eighth week of inspiratory muscle training, and 3) at the end of the training (twelfth) week. During inspiratory muscle training, individuals will attend on Hospital de Clinicas de Porto Alegre, once a week, to the supervision of the way the exercise is being performed. Furthermore, it will be set to load on the PowerBreathe ® device for the following week.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes;
* 30 years and older;
* HbA1c from 7,5 to 10%.

Exclusion Criteria:

* Pregnant women;
* Pulmonary disease (chronic obstructive pulmonary disease, exercise-induced asthma, idiopathic pulmonary fibrosis, sarcoidosis and lung neoplasms);
* Neuromuscular disease;
* Body mass index > 35 kg/m²;
* Individuals who perform physical exercise more than twice a week;
* Current smoking.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin in 8 weeks | Evaluated in 8 weeks of inspiratory muscle training
  Glycated hemoglobin concentration after 8 weeks of inspiratory muscle training
Glycated hemoglobin in 12 weeks | Evaluated in 12 weeks of inspiratory muscle training
  Glycated hemoglobin concentration after 12 weeks of inspiratory muscle training

SECONDARY OUTCOMES:
Glucose in 8 weeks | Evaluated in 8 weeks of inspiratory muscle training
  Fasting plasma glucose concentration after 8 weeks of inspiratory muscle training.
Glucose in 12 weeks | Evaluated in 12 weeks of inspiratory muscle training
  Fasting plasma glucose concentration after 12 weeks of inspiratory muscle training.
Respiratory muscle strength in 8 weeks | Evaluated in 8 weeks of inspiratory muscle training
  Maximum respiratory muscle strength after 8 weeks of inspiratory muscle training, through the measurement of the maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP).
Respiratory muscle strength in 12 weeks | Evaluated in 12 weeks of inspiratory muscle training
  Maximum respiratory muscle strength after 12 weeks of inspiratory muscle training, through the measurement of the maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP).
Ventilatory muscle resistance | Evaluated in 12 weeks of inspiratory muscle training
  Muscular endurance ventilatory after 12 weeks of inspiratory muscle training, through analysis of the MIP.
Lung functions | Evaluated in 12 weeks of inspiratory muscle training
  Capacity and volumes lung after 12 weeks of inspiratory muscle training.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz D'Agord Schaan, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pinto MB, Bock PM, Schein ASO, Portes J, Monteiro RB, Schaan BD. Inspiratory Muscle Training on Glucose Control in Diabetes: A Randomized Clinical Trial. Int J Sport Nutr Exerc Metab. 2021 Jan 1;31(1):21-31. doi: 10.1123/ijsnem.2020-0175. Epub 2020 Nov 27. PMID 33248438